CLINICAL TRIAL: NCT04617522
Title: A Phase 1, Open-Label, Dose-Escalation Study to Determine an Appropriate Starting Dose of Sacituzumab Govitecan in Subjects With Advanced or Metastatic Solid Tumor and Moderate Liver Impairment
Brief Title: Study of Sacituzumab Govitecan in Participants With Advanced or Metastatic Solid Tumor and Moderate Liver Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-15; 2022-501508-82 (Other: EU CT Number)
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced or Metastatic Solid Tumor; Liver Failure
MeSH Terms: conditions — Neoplasm Metastasis; Liver Failure | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Advanced or Metastatic Solid Tumor and Moderate Liver Impairment (Experimental): Participants with advanced solid tumor and moderate hepatic impairment will receive an escalating dose of sacituzumab govitecan-hziy on Days 1 and 8. The dose-escalation plan will start at 5 mg/kg and escalate to 7.5 mg/kg, and finally 10 mg/kg, if deemed to be safe. At the completion of study treatment, participants who are deriving benefit from sacituzumab govitecan-hziy may continue to receive treatment in a Gilead sponsored rollover study (IMMU-132-14; NCT04319198).
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Advanced or Metastatic Solid Tumor and Normal Liver function (Experimental): Participants with advanced or metastatic solid tumor and normal hepatic function will receive sacituzumab govitecan-hziy 10 mg/kg on Days 1 and 8. At the completion of study treatment, participants who are deriving benefit from sacituzumab govitecan-hziy may continue to receive treatment in a Gilead sponsored rollover study (IMMU-132-14; NCT04319198).
  Interventions: Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; GS-0132

SUMMARY:
The goals of this clinical study are to learn more about the safety and dosing of the study drug, sacituzumab govitecan-hziy, in participants with solid tumors and moderate liver problems.

ELIGIBILITY:
Key Inclusion Criteria for all Individuals:

* Histologically confirmed advanced or metastatic solid tumor that is measurable or nonmeasurable.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥1,500/mm^3, and platelets ≥ 100,000/ μL).
* Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation.

Key Inclusion Criteria for Individuals with Normal Hepatic Function:

* Normal hepatic function (total bilirubin ≤ ULN and aspartate aminotransferase (AST) ≤ 3.0× ULN).

Key Inclusion Criteria for Individuals with Moderate Hepatic Function:

* Moderate hepatic impairment (1.5 × ULN < total bilirubin ≤ 3.0 × ULN and any level of AST).
* For individuals with hepatic encephalopathy, the condition does not, in the Investigator's opinion, interfere with the individual's ability to provide an appropriate informed consent.

Key Exclusion Criteria for all Individuals:

* Have poor venous access.
* Donated or lost 500mL or more of blood volume (including plasmapheresis) to plans to donate during the study.
* Have had a prior anticancer biologic agent within 4 weeks prior to Day 1 or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Day 1 and who have not recovered (i.e., ≤ Grade 1) from adverse events (AEs) at the time of study entry. Individuals participating in observational studies are eligible.
* Had prior treatment with irinotecan within 4 weeks prior to Day 1.
* Have not recovered (i.e., ≤ Grade 1) from AEs due to a previously administered agent.
* Have an active second malignancy.
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Individuals with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking < 20 mg/day of prednisone or its equivalent. All individuals with carcinomatous meningitis are excluded regardless of clinical stability.
* Have history of cardiac disease.
* Have active chronic inflammatory bowel disease (ulcerative colitis or Crohn's disease) or gastrointestinal (GI) perforation within 6 months of enrollment.
* Have active serious infection (Contact medical monitor for clarification).
* High-dose systemic corticosteroids (≥20 mg of prednisone or its equivalent) are not allowed within 2 weeks of Check-In. However, inhaled, intranasal, intra-articular, and topical steroids are allowed.
* Use of strong inhibitor or inducer of UGT1A1.
* Have a known history of Gilbert's disease.

Key Exclusion Criteria for Individuals with Normal Hepatic Impairment:

* Must have pre-existing condition interfering with hepatic and/or renal function that could interfere with the metabolism and/or excretion of the study drug.

Key Exclusion Criteria for Individuals with Moderate Hepatic Impairment:

* Had a significant clinical exacerbation of liver disease symptoms within the 2-week period before administration of study drug (i.e., abdominal pain, nausea, vomiting, anorexia, or fever).
* Had clinically demonstrable, tense ascites.
* Had evidence of acute viral hepatitis within 1 month prior to administration of study drug.
* Have evidence of hepatorenal syndrome.
* Individuals with transjugular intrahepatic portosystemic shunt (TIPS) placement.
* Have active Stage 3 or 4 encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants experiencing Treatment Emergent Adverse Events (TEAEs) and Serious AEs | First dose date up to Day 38
Percentage of Participants Experiencing Any Dose Limiting Toxicities (DLTs) | Up to Day 22 (for participants receiving SG on Day 1); Up to Day 28 (for participants receiving SG on Day 8)
Percentage of Participants Experiencing Any Clinically Significant Laboratory Abnormalities | First dose date up to Day 38
Pharmacokinetic (PK) Parameter: Cmax of Free SN-38 and Sacituzumab Govitecan-hziy | Days 1 and 8
  Cmax will be determined for 2 analytes: Free SN-38 and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. Cmax is defined as the maximum observed concentration obtained directly from the observed concentration-time data.
PK Parameter: AUC 0-168 of Free SN-38 and Sacituzumab Govitecan-hziy | Days 1 and 8
  AUC 0-168 will be determined for 2 analytes: Free SN-38 and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. AUC0-168 is defined as area under the serum concentration-time curve from time 0 to 168 hours.
Percentage of Participants who Develop Anti-Sacituzumab Govitecan-hziy Antibodies | Day 1 (Predose) and Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- United States (8):
  - Pacific Shores Medical Group, Long Beach, California
  - Christiana Care Health Services, Newark, Delaware
  - University of Maryland, Baltimore, Maryland
  - NEXT Austin, Austin, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - NEXT Oncology, San Antonio, Texas
- France (3):
  - Institut Bergonie Medical Oncology, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut de Cancerologie de l'Ouest (ICO) - Saint-Herblain, Saint-Herblain
- Spain (2):
  - Institut Català d'Oncologia - L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardillo TM, Govindan SV, Sharkey RM, Trisal P, Goldenberg DM. Humanized anti-Trop-2 IgG-SN-38 conjugate for effective treatment of diverse epithelial cancers: preclinical studies in human cancer xenograft models and monkeys. Clin Cancer Res. 2011 May 15;17(10):3157-69. doi: 10.1158/1078-0432.CCR-10-2939. Epub 2011 Mar 3. PMID 21372224
- [Background] Cardillo TM, Govindan SV, Sharkey RM, Trisal P, Arrojo R, Liu D, Rossi EA, Chang CH, Goldenberg DM. Sacituzumab Govitecan (IMMU-132), an Anti-Trop-2/SN-38 Antibody-Drug Conjugate: Characterization and Efficacy in Pancreatic, Gastric, and Other Cancers. Bioconjug Chem. 2015 May 20;26(5):919-31. doi: 10.1021/acs.bioconjchem.5b00223. Epub 2015 May 8. PMID 25915780
- [Background] Cardillo TM, Sharkey RM, Rossi DL, Arrojo R, Mostafa AA, Goldenberg DM. Synthetic Lethality Exploitation by an Anti-Trop-2-SN-38 Antibody-Drug Conjugate, IMMU-132, Plus PARP Inhibitors in BRCA1/2-wild-type Triple-Negative Breast Cancer. Clin Cancer Res. 2017 Jul 1;23(13):3405-3415. doi: 10.1158/1078-0432.CCR-16-2401. Epub 2017 Jan 9. PMID 28069724
- [Background] Goldenberg DM, Cardillo TM, Govindan SV, Rossi EA, Sharkey RM. Trop-2 is a novel target for solid cancer therapy with sacituzumab govitecan (IMMU-132), an antibody-drug conjugate (ADC). Oncotarget. 2015 Sep 8;6(26):22496-512. doi: 10.18632/oncotarget.4318. Erratum In: Oncotarget. 2020 Mar 10;11(10):942. doi: 10.18632/oncotarget.27512. PMID 26101915
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Derived] Kwapisz D. Sacituzumab Govitecan-hziy in Breast Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):279-285. doi: 10.1097/COC.0000000000000919. Epub 2022 May 12. PMID 35728046
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=IMMU-132-15